CLINICAL TRIAL: NCT07317271
Title: Virtual Reality-Enhanced Progressive Muscle Relaxation for Symptom Management in Burn Survivors
Brief Title: VR-PMR for Post-Burn Symptoms
Acronym: VIBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00488719
Record Dates: First submitted 2025-12-10; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Burn; Chronic Pain Following Thermal Burn Injury; Non-Pharmacological Interventions; Virtual Reality; Sleep Disturbance; Anxiety; Depressive Symptoms; Fatigue Symptom; Pruritus; Burn Injury; Progressive Muscle Relaxation
Keywords: Virtual Reality; Burn Survivors; Progressive Muscle Relaxation; Chronic Symptom Management; Pain; Itch; Sleep; Fatigue; Burns; Burn Injury
MeSH Terms: conditions — Burns; Parasomnias; Anxiety Disorders; Depression; Fatigue; Pruritus; Pain

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, two-period, two-treatment crossover interventional model to compare the effects of standard PMR with VR-enhanced PMR (VR-PMR). Each participant receives both interventions in a randomized sequence, allowing each individual to serve as the individual's own control. This design improves statistical power with a relatively small sample and minimizes confounding from inter-individual differences such as burn severity, baseline symptom levels, and psychosocial characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-PMR (Experimental)
  Interventions: Behavioral: Virtual Reality-Enhanced Progressive Muscle Relaxation
- PMR (Active Comparator)
  Interventions: Behavioral: Standard Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Virtual Reality-Enhanced Progressive Muscle Relaxation — The VR-PMR intervention is a self-administered 20-minute session, conducted for 3 consecutive days, one hour before bedtime. PMR, participants will tighten and relax specific muscle groups in sequence from the upper body to the lower body then vice versa. While taking deep breaths inhaling through the nose and exhaling through the mouth, patients will be asked to first tense a muscle tightly and hold for slow count of 5 seconds and then relax quickly and completely for 10 seconds until all the tightness and pain flow out of the muscles. During PMR, participants will be immersed in a relaxing, nature-based VR environment. The VR component will use the Quest 3 Headset. Participants will be immersed in a virtual nature walk with accompanying relaxing music and nature sounds. Participants will be given a choice of three 360 nature walk videos set in forests or a beach. Audio instructions for PMR will play over the video's audio. Participants will use the participant's own smartphone.
  Arms: VR-PMR
Behavioral: Standard Progressive Muscle Relaxation — Standard progressive muscle relaxation (PMR) therapy delivered via audio-recorded guides. For PMR, participants will tighten and relax specific muscle groups in sequence from the upper body to the lower body then vice versa. While taking deep breaths inhaling the nose and exhaling through the mouth, patients will be asked to first tense a muscle tightly and hold for slow count of 5 seconds and then relax quickly and completely for 10 seconds until all the tightness and pain flow out of the muscles.
  Arms: PMR

SUMMARY:
The goal of this clinical trial is to learn whether progressive muscle relaxation (PMR), delivered either alone or enhanced with virtual reality (VR), can help treat chronic symptom, such as pain, itch, anxiety, sleep disturbances, and fatigue, in adult burn survivors.

The main questions it aims to answer are:

* Does VR-enhanced PMR (VR-PMR) reduce chronic pain, anxiety, itch, sleep disturbances, and fatigue more effectively than standard PMR?
* Is VR-PMR a feasible and acceptable self-administered home-based intervention for burn survivors?

Researchers will compare two self-administered intervention conditions, VR-enhanced PMR and standard PMR, using a randomized to sequence crossover design to see if VR technology enhances the therapeutic effects of PMR on chronic symptom management in burn survivors.

Participants will:

* Complete home-based sessions of VR-enhanced PMR
* Complete home-based sessions of standard PMR
* Report symptoms such as pain, itch, anxiety, sleep disturbances, and fatigue throughout the study
* Use VR equipment provided for the intervention period (during the VR-PMR arm)

DETAILED DESCRIPTION:
Serious burn injuries are a devastating form of trauma, often resulting in long-term physical and psychological challenges. Burn survivors experience a host of burdensome and co-occurring chronic symptoms post-burn injury that affect quality of life and recovery. Among the most prevalent are pain, pruritis (itch), anxiety, sleep disturbances, and fatigue. Despite a decrease in intensity over time, these symptoms often persist well-beyond the initial burn injury and negatively impact recovery, activities of daily living, social participation, and quality of life. Research indicates that these symptoms often co-occur and demonstrate bidirectional relationships. For instance, pain and itch can contribute to sleep disturbances, while anxiety and fatigue can worsen overall itch and pain perception. A reciprocal relationship between sleep and pain after burn injuries has been demonstrated in a number of studies suggesting that pain contributes to poor sleep, and that disruptions in sleep are associated with increased pain and increased use of analgesics.

Pharmacologic interventions for these symptoms, such as the use of opioids or sedatives, can have adverse effects, including dependence, side effects, and inadequate long-term relief. Given the limitations of pharmacologic interventions, non-pharmacologic therapies, such as cognitive-behavioral therapy (CBT), mindfulness, and relaxation techniques, have gained recognition as effective strategies for symptom management in this population. However, CBT, often regarded as the gold standard intervention for improving sleep and pain, has its own barriers, including the need for trained professionals, high costs, and challenges related to patient adherence. These barriers underscore the need for cost-effective, accessible, and effective self-administered approaches that can be easily integrated into everyday life of burn survivors.

Progressive muscle relaxation (PMR) is a well-established mind-body relaxation technique that has been shown to reduce stress, anxiety, pain, and itch, and improve sleep by systematically tensing and relaxing different muscle groups. Recent advancements in virtual reality (VR) technology present an opportunity to enhance the delivery of PMR by creating immersive environments that promote relaxation and improve therapeutic outcomes. VR has previously been used to enhance existing therapies to help improve engagement and therapeutic by providing an immersive environment that complements the therapy. It has been shown to provide pain relief and reduce anxiety in various clinical settings and populations, such as burn care, procedural pain, and chronic pain management. VR is hypothesized to facilitate a more realistic and relaxing sensory experience and has the potential to amplify the effects of PMR by providing additional relaxing auditory and visual stimuli.

This study would leverage novel VR technology to enhance a well-established mind-body intervention, PMR, to support symptom management in a burn population. While the combination of VR and PMR has been explored in a variety of pain populations, its effect on chronic pain, anxiety, itch, sleep, and fatigue have yet to be explored in a burn population. Therefore, this proposed study seeks to evaluate the use of a novel self-administered VR-enhanced PMR (VR-PMR) therapy delivered at-home for symptom management in burn survivors. The aims for this study are as follows:

Aim 1. Determine the feasibility of an at-home, self-administered VR-enhanced PMR (VR-PMR) and PMR intervention in burn survivors.

Aim 1a. Recruitment, enrollment, retention rates, and intervention adherence of participants will be recorded and used to help determine feasibility of the VR-PMR intervention.

Aim 1b. Usability of VR-PMR intervention will be measured with surveys and open-ended prompts for additional qualitative feedback.

Aim 2. Evaluate the preliminary efficacy of VR-PMR and standard PMR interventions on symptom outcomes, including pain severity, itch severity, anxiety, sleep quality, and fatigue, using a within-subject crossover design.

Aim 2a. Compare changes in symptom outcomes across both intervention phases to identify any differential effects.

Aim 2b. Assess the presence of any carryover effects between intervention phases and the potential impact on outcome measures.

ELIGIBILITY:
Inclusion criteria are:

* ≥18 years old;
* sustained a burn injury in the last 6 months or longer;
* Score high on at least one of the following: Insomnia severity index (ISI) score of ≥8, Brief Pain Inventory Short Form (BPI-SF) Pain severity score of ≥3, or PROMIS Itch Severity of ≥55;
* own a smartphone or computer with reliable internet connection for online visits and survey completion;
* able to comfortably wear goggles or headsets on face as determined by self-report.

Exclusion criteria:

* Cognitive impairment (Mini Mental Status Exam (MMSE) < 25);
* history of motion sickness, photosensitivity, photoinduced seizures, and claustrophobia as determined by self-report;
* uncorrected visual or hearing impairments as determined by self-report;
* non-English speaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity as assessed by the the Numeric Rating Scale (NRS). | pre intervention and post VR-PMR intervention (3 weeks)
  Pain will be measured using the the Numeric Rating Scale (NRS). Scale range 0-10, higher score worse pain severity.
Itch Intensity as assessed by the the Numeric Rating Scale (NRS) | pre intervention and post VR-PMR intervention (3 weeks)
  Itch intensity pre- and post-intervention will be measured using the the Numeric Rating Scale (NRS). Scale range 0-10, higher score worse itch severity.
Anxiety as assessed by the Numeric Rating Scale | Pre intervention, post VR-PMR intervention (3 weeks)
  Anxiety severity pre- and post-intervention will be measured using the Numeric Rating Scale. Total score range from 0-10 with higher scores indicating worse anxiety.

SECONDARY OUTCOMES:
Quality of Life (Burn Specific Health Scale Brief) | pre intervention and post intervention (3 weeks)
  The Burn Specific Health Scale Brief (BSHS-B) will assess quality of life pre- and post-intervention. The BSHS-B consists of 40-items with 9 subscales that measure physical and psychosocial aspects of burn recovery. Total score range 0-160 (sum of score for all items) higher score suggests better quality of life.
Sleep Disturbances as assessed by the PROMIS Sleep Disturbance Scale | pre intervention and post intervention (3 weeks)
  The PROMIS Sleep Disturbance scale will be used to measure pre- and post-intervention sleep quality. T score mean = 50, SD = 10 Higher scores indicate worse symptoms.
Total Sleep Time (TST) | pre intervention and post intervention (3 weeks)
  Total sleep time (minutes) derived from actigraphy and sleep diary data.
Wake After Sleep Onset (WASO) | pre intervention and post intervention (3 weeks)
  Derived from actigraphy and sleep diary data.
Sleep Latency | pre intervention and post intervention (3 weeks)
  Derived from actigraphy and sleep diary data. Amount of time measured in minutes it takes to fall asleep.
Sleep Efficiency | pre intervention and post intervention (3 weeks)
  Derived from actigraphy and sleep diary data. Percentage total sleep time divided by time in bed.
Fatigue as assessed by the Multidimensional Fatigue Inventory | pre intervention and post intervention (3 weeks)
  Fatigue will be measured using the Multidimensional Fatigue Inventory (MFI) at baseline and at the end of the PMR sessions. The MFI is a 20-item scale designed to evaluate 5 dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Scores on each subscale range 4-20. Total score range 20 to 100; higher the score worse fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Sheera Lerman Zohar, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States